CLINICAL TRIAL: NCT00304330
Title: Emergence of Gram-negative Resistance in Blood Culture Isolates of Solid-organ Transplant Recipients; a Comparative Study With a Non-transplant Population
Brief Title: Emergence of Gram-negative Resistance in Blood Culture Isolates of Solid-organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 0602123; NCT00332423 (obsolete NCT alias)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Gram Negative Infection
Keywords: gram negative infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The information collected will provide insight in to the epidemiology of antibiotic resistance in a transplant compared to a non-transplant population. Data is needed regarding the date of admission, date of bloodstream infection and location of ward/ICU so trends in the emergence of resistance and antibiotic usage can be detected.

DETAILED DESCRIPTION:
We need to collect details on the demographics (age, sex etc), underlying conditions, transplant types and immunosuppression, in-hospital antibiotic management and clinical outcomes so that the effect of antibiotic resistance on patient outcome can be measured. We also need to collect microbiology and pathology data to determine the antibiotic susceptibility profile of the involved organisms. The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, prophylactic antimicrobials, physical exam findings, laboratory and radiographical data, empiric antimicrobial usage, microbiological data and resistance patterns, choice of antibiotic once organism identified, suspected source of infection, microbiological and clinical outcomes, laboratory results, demographic information, medications, gender, weight, ethnicity, and past medical history

ELIGIBILITY:
Inclusion Criteria:

* All patients with a positive blood culture isolate growing a gram-negative organism will be included from 1996 - 2005

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: gram negative organisms
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2006-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States